CLINICAL TRIAL: NCT06417320
Title: Effect of Sodium-glucose Cotransporter-2 Inhibitors (SGLT-2i) on Proteinuria in Nephrotic Children Older Than 10 Years
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.22.11.2207
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Nephrotic Syndrome in Children
MeSH Terms: interventions — Angiotensin-Converting Enzyme Inhibitors; Captopril; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 (ACEI group)
  Interventions: Drug: ACEI, SGLT-2i
- Group 2 (Active Comparator): Group 2 (combined ACEI and SGLT-2i group)
  Interventions: Drug: ACEI, SGLT-2i

INTERVENTIONS:
Drug: ACEI, SGLT-2i — Group 1 (ACEI group) will receive a single dose of oral ACE inhibitors tablets per day (0.2-0.6mg) /kg/ day)
  ❖ Group 2 (combined ACEI and SGLT-2inhibitrs group) patients on a single dose of oral ACE inhibitors tablets per day (0.2-0.6mg /kg/ day) presenting with persistent nephrotic range proteinuria will add a single dose of oral SGLT-2 inhibitors tablets 5mg per day (weight≤30kg) or 10mg per day (weight >30kg)
  Other Names: Captopril, forxiga

SUMMARY:
The goal of this clinical trial is to evaluate the effect of ACE inhibitors and SGLT-2 inhibitors on:

1. Proteinuria
2. Renal survival indices

DETAILED DESCRIPTION:
This is a randomized, double blind study. Patients are randomized to receive oral ACE inhibitors or combined ACEI and SGLT-2inhibitrs once daily for12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 and 18 years old,
* Nephrotic resistant patients,
* No history of diabetes,
* Estimated GFR≥60ml/min/1.73m2, will be evaluated by Schwartz formula,
* Caregivers' acceptance to be enrolled in the study.

Exclusion Criteria:

* Uncontrolled urinary tract infection at screening,
* Blood pressure is less than 5th percentile of the same gender, age, height,
* At risk of dehydration or volume depletion,
* Evidence of liver disease: defined by serum levels of alanine transaminase or aspartate transaminase >2 times the upper limit of normal during screening,
* History of organ transplantation, cancer, liver disease,
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Protein free period, eGFR | 12 weeks following end of treatment
  Protein free period by test strips (dipstick) and microscopy, urine protein/creatinine ratio and Estimated GFR will be evaluated by Schwartz formula

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Refaey, MBBCh,MSc,MD, Study Director — Mansoura University-Faculty of Medicine-Pediatric
Locations (1):
- Mansoura University Children's Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing of study protocol
Supporting Information: Study Protocol
Time Frame: 1year
Access Criteria: any one